CLINICAL TRIAL: NCT07262424
Title: The Influence of Instructor-centered Versus Learner-centered Debriefing on Clinical Judgment in Nursing Students: A Mixed-methods Experimental Study Protocol.
Brief Title: Debriefing Styles and Clinical Judgment in Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Aleix Lopez Oganissian, MsC, PhdCandidate, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LCTandICTDebriefing&ClinJudge
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Simulation Based Learning; Nursing Education; Debriefing Method
Keywords: Clinical Judgment; Learner-Centered Teaching; Instructor-Centered Teaching; Mixed-Methods Study; Debriefing; Nursing Education; Simulation; Randomized Controlled Trial; Undergraduate Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learner-Centered Debriefing (LCT) (Experimental): Participants in this group will receive a debriefing guided by a learner-centered (LCT) style, where learning is a dynamic process of meaning-making, and both learners and instructors collaborate in the co-construction of knowledge, skills, and attitudes.
  Interventions: Behavioral: Learner-Centered Debriefing
- Instructor-Centered Debriefing (ICT) (Active Comparator): Participants in this group will receive a debriefing guided by an instructor-centered (ICT) style, which prioritizes the efficient transfer of information from instructors (who control the learning environments) to learners.
  Interventions: Behavioral: Instructor-Centered Debriefing

INTERVENTIONS:
Behavioral: Learner-Centered Debriefing — Two 2-hour simulation sessions followed by a learner-centered debriefing conducted by a trained facilitator. This style emphasizes guided reflection and co-construction of knowledge.
  Arms: Learner-Centered Debriefing (LCT)
Behavioral: Instructor-Centered Debriefing — Two 2-hour simulation sessions followed by an instructor-centered debriefing conducted by a trained facilitator. This style is the standard practice at the institution and focuses on direct feedback and information transfer from the instructor.
  Arms: Instructor-Centered Debriefing (ICT)

SUMMARY:
Simulation is a cornerstone of health sciences education, with debriefing being its most critical component for fostering clinical skills. While various debriefing styles exist, there is limited evidence comparing the effectiveness of instructor-centered (ICT) versus learner-centered (LCT) approaches, specifically on the development of clinical judgment in nursing students.

DETAILED DESCRIPTION:
Several studies suggest a general preference for a Learner-Centered (LCT) style during simulation debriefing. However, existing literature and expert opinion often recommend an Instructor-Centered (ICT) style for novice learners or in time-limited situations. It is critical to note that these recommendations are not consistently based on robust scientific evidence, highlighting a significant gap in nursing education research. This study is designed to address this gap by systematically evaluating the impact of ICT versus LCT debriefing on the acquisition of clinical judgment in undergraduate nursing students-a cornerstone competency for professional practice.

The study's central hypothesis is: "The debriefing style, whether instructor-centered (ICT) or learner-centered (LCT), differently impacts students' learning process in clinical judgment."

To test this hypothesis, the study employs a mixed-methods sequential explanatory design. The initial quantitative phase consists of a randomized controlled trial to determine the effect of the two debriefing styles. This will be followed by a qualitative phase, utilizing focus groups, to explore the students' perceptions and experiences, thereby providing a deeper, contextual explanation for the quantitative findings.

To ensure the integrity of the intervention, methodological fidelity will be rigorously monitored. The distinction between the ICT and LCT styles will be verified through objective measures, including the analysis of faculty-to-student talk-time ratios and the mapping of conversation patterns (sociograms) during debriefing sessions. This ensures that the observed differences in learning can be confidently attributed to the assigned debriefing style. The integration of both quantitative and qualitative data will yield a comprehensive understanding of how different pedagogical approaches in simulation debriefing influence the complex process of clinical judgment development.

ELIGIBILITY:
Inclusion Criteria:

-Students enrolled in the Basic Simulation Labs 2 (LBS2) course as part of their program.

Exclusion Criteria:

* Students who cannot participate in all phases of the study.
* Students who do not provide informed consent.
* Students who are repeating the course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Judgment Assessed by the Lasater Clinical Judgment Rubric (LCJR) | Assessed at two time points: at Baseline (measurement taken during the first-term practical exam, prior to the intervention) and Post-Intervention (measurement taken during the final practical exam, approximately 3 months after the baseline assessment).
  Assessment is performed using the Lasater Clinical Judgment Rubric (LCJR), a validated 11-item tool. During a standardized practical exam (OSCE), trained evaluators will use novel structured checklists developed by the investigators for this study. A unique checklist has been specifically tailored for each OSCE scenario, designed to operationalize the LCJR by mapping observable student behaviors directly to its scoring criteria. Each item is rated on a 4-point scale (1=beginning to 4=exemplary), yielding a total score from 11 to 44. A higher score indicates a more developed level of clinical judgment. For statistical analysis, the raw score will be transformed to a 0-10 scale.

SECONDARY OUTCOMES:
Student Perceptions of the Learning Experience Assessed by Focus Group Topic Guide | Up to 3 weeks after the final simulation session.
  Perceptions and experiences of students and faculty regarding how different debriefing styles influenced the learning of clinical judgment will be explored through semi-structured focus groups. Data collection will be guided by a Focus Group Topic Guide designed to elicit feedback on the debriefing style, application of theoretical concepts, and the learning experience. The metric for assessment is qualitative, consisting of the identification and categorization of recurring themes and sub-themes derived from the thematic analysis of transcribed discussions.

CONTACTS AND LOCATIONS:
Locations (1):
- International University of Catalonia, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Background] Eppich W, Cheng A. Promoting Excellence and Reflective Learning in Simulation (PEARLS): development and rationale for a blended approach to health care simulation debriefing. Simul Healthc. 2015 Apr;10(2):106-15. doi: 10.1097/SIH.0000000000000072. PMID 25710312
- [Background] Roman-Cereto M, Garcia-Mayor S, Kaknani-Uttumchandani S, Garcia-Gamez M, Leon-Campos A, Fernandez-Ordonez E, Ruiz-Garcia ML, Marti-Garcia C, Lopez-Leiva I, Lasater K, Morales-Asencio JM. Cultural adaptation and validation of the Lasater Clinical Judgment Rubric in nursing students in Spain. Nurse Educ Today. 2018 May;64:71-78. doi: 10.1016/j.nedt.2018.02.002. Epub 2018 Feb 9. PMID 29459195
- [Background] Cheng A, Morse KJ, Rudolph J, Arab AA, Runnacles J, Eppich W. Learner-Centered Debriefing for Health Care Simulation Education: Lessons for Faculty Development. Simul Healthc. 2016 Feb;11(1):32-40. doi: 10.1097/SIH.0000000000000136. PMID 26836466